CLINICAL TRIAL: NCT03388463
Title: The Effectiveness of Standard Single Dose Omeprazole Versus High Dose Continuous Infusion in High-risk Critically Ill Patients.
Brief Title: Single Dose Omeprazole Versus High Dose in High-risk Critically Ill Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Assistant Professor in anaesthesia, intensive care, and pain medicine., Menoufia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MenoufiaU2016/2ICU
Record Dates: First submitted 2017-12-24; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omeprazole group (Active Comparator): Patients received intravenous bolus of 80 mg omeprazole followed by 8mg/h infusion for the whole period of ICU stay.
  Interventions: Drug: Omeprazole
- Placebo group (Placebo Comparator): Patients received intravenous omeprazole 40mg bolus dose once daily followed by normal saline infusion.
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Omeprazole — Omeprazole 80 mg continues infusion
  Other Names: Omeprazole continues infusion
  Arms: Omeprazole group
Drug: Placebo group — Omeprazole 40 mg single daily dose.
  Other Names: Placebo for infusion
  Arms: Placebo group

SUMMARY:
Upper gastrointestinal (GIT) bleeding is common in high risk critically ill patients. Hyperacidity has been identified as one of the main reasons for bleeding.1 2 Antacids with different treatment modalities have been studied to establish the best regimen for prophylaxis against bleeding.3 4 Proton pump inhibitors (PPI) are the most common drugs used in the medical field as antacids. The present study was carried out to investigate the beneficial effects of high dose omeprazole versus standard low dose as a prophylaxis against upper GIT bleeding in high risk critically ill patients.

DETAILED DESCRIPTION:
A hundred and ten high risk critically ill patients were divided into two groups, fify five patients each. Group A received intravenous (IV) omeprazole 40mg bolus dose once daily followed by normal saline infusion. Group B received IV bolus of 80 mg omeprazole followed by 8mg/h infusion. The treatment was for the whole period of ICU stay. Gastric pH, residual gastric volume, signs of significant upper GIT bleeding, ICU stay Hb, number of ventilator free days, ICU stay haemoglobin (Hb), number of red cell units transfused in ICU, ICU stay, and numbers of ICU survivors were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients were identified as high risk patients. Patients with nasogastric tube inserted as part of their medical care were included in the study.

Exclusion Criteria:

* Patients admitted because of upper gastrointestinal bleeding, patients who were not scheduled for early enteral nutrition during the first 24 hours of intensive care unit (ICU) admission, patients with bleeding disorders, renal replacement therapy, history of gastric ulcer, gastric surgery, and the use of gastric antacids before ICU admission.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
Significant upper gastrointestinal bleeding | 20 days during ICU stay.
  Vomiting of fresh blood, melena, or haematemesis.